CLINICAL TRIAL: NCT06764199
Title: The Effect of an Acceptance and Commitment Therapy-Based Psychoeducation Program Applied to Individuals with Chronic Mental Disorders on Patients' Perceptions of Stigmatization, Functionality, and Quality of Life Levels
Brief Title: The Effect of an Acceptance and Commitment Therapy-Based Psychoeducation Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ceylan Aksoy, Principal Investigator, Ataturk University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/618
Record Dates: First submitted 2024-12-19; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Chronic Mental Disorders
MeSH Terms: interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention Group (Experimental): Acceptance and Commitment Therapy will be applied.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Participant Group (No Intervention): Only data collection was carried out. No attempt was made by the researcher during the study.
- Control Group (No Intervention): Only data collection was carried out. No attempt was made by the researcher during the study.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Acceptance and Commitment Therapy (ACT), a relatively new psychotherapy, incorporates psychopathological hypotheses and interventions based on contextual behavioral sciences and Relational Frame Theory.
  Arms: Intervention Group

SUMMARY:
The concept of mental disorders is defined as health conditions characterized by various changes in individuals' emotions, thoughts, behaviors, and cognitive processes. The most significant feature of mental disorders is the frequent recurrence and persistence of psychiatric symptoms. Due to their widespread prevalence in society and their substantial contribution to disability, mental disorders are among the groups of diseases requiring early intervention, particularly due to their chronic nature. Chronic mental disorders are associated with hallucinations, delusions, self-stigmatization, and reduced quality of life. Chronic conditions such as schizophrenia, bipolar disorder, and schizoaffective disorder are reported in the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) to be linked with impairments in occupational and social functionality.

In the literature, these chronic mental disorders are often referred to as "severe," "persistent," or "serious" mental illnesses due to their destructive effects on cognitive, executive, and social skills. Chronic mental disorders, which cause significant disability, are considered a public health issue. Even when the symptoms of diseases such as schizophrenia, bipolar disorder, and schizoaffective disorder are treated, the resulting functional impairments often persist for an extended period, posing a significant burden on both individuals and society. Studies conducted in hospital and community mental health centers have indicated that individuals diagnosed with schizophrenia and bipolar disorder experience impairments in social functioning and significant disabilities.

Research highlights various challenges faced by individuals with chronic mental disorders, such as deterioration in social relationships, stigmatization, lack of motivation, insufficient self-care, and challenges in daily living skills like financial management, communication, and shopping. Another critical issue in individuals with chronic mental disorders is self-stigmatization, which is closely related to social disadvantage and functionality. Studies examining the self-stigmatization levels of these individuals have reported an increase in such behaviors, identifying self-stigma as a significant global concern in the literature.

Consequently, it is evident that psychosocial interventions addressing functionality, insight, and self-stigmatization levels, which are thought to be interrelated, should be prioritized for individuals with chronic mental disorders. Addressing these issues underscores the importance of psychiatric rehabilitation activities designed for this population.

While pharmacotherapy is the first choice in the treatment of chronic mental disorders, research indicates that medications alone do not achieve clinically significant improvements in negative and cognitive symptoms, nor do they produce the desired outcomes in functionality. Current guidelines emphasize that the inclusion of psychosocial interventions alongside pharmacotherapy can yield more favorable outcomes in the prognosis of psychotic disorders. Treatment of chronic mental disorders should not only focus on mitigating psychotic symptoms but also aim to improve quality of life, social, and occupational functioning.

Acceptance and Commitment Therapy (ACT), a relatively new psychotherapy, incorporates psychopathological hypotheses and interventions grounded in contextual behavioral sciences and Relational Frame Theory. Limited studies have shown that ACT applied to patients with psychosis reduces levels of depression and anxiety, enhances psychological resilience, facilitates independent daily living, and thereby improves functionality. In light of these findings, psychosocial interventions for individuals with chronic mental disorders are deemed highly valuable. It is anticipated that ACT applied to these individuals may positively alter the course of the illness, reduce self-stigmatization and internalized shame, contribute to improved functionality, and ultimately enhance quality of life. Conducting research to explore the significance and effectiveness of these interventions is of utmost importance.

ELIGIBILITY:
Inclusion Criteria:

* Being registered with a Community Mental Health Center (CMHC).
* Providing consent to participate in the study, either personally or through a legal guardian.
* Being between the ages of 18 and 65. Being literate.
* According to the treatment team and records, having been in a stable condition for at least six months.

Exclusion Criteria:

* Being under 18 years of age.
* Presence of an organic psychotic disorder.
* Experiencing an episode during the intervention process.
* Refusing to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Self-Stigma Scale | 1 year
  It was developed to accurately assess self-stigma in individuals with mental illnesses by ensuring that patients understand the questions and that the items reflect the stigma they experience within their cultural context. The scale consists of 17 items, with no reverse-scored items. Responses to each item are rated on a 5-point Likert scale: 1 = strongly disagree, 2 = somewhat disagree, 3 = moderately agree, 4 = generally agree, and 5 = completely agree. Higher scores indicate higher levels of self-stigma. The scale's Cronbach's alpha correlation coefficient is 0.93, indicating high reliability.

SECONDARY OUTCOMES:
Social Functioning Assessment Scale | 1 year
  It is a 19-item Likert-type scale developed for schizophrenia patients. Each item is in the range of 1-3 points. It is seen that the scale consists of four factors as interpersonal relations and entertainment, self-care, independent living skills and working life. The score that can be obtained from the scale is in the range of 19-57, and a high score from the scale means that the individual has a high level of social functionality.
Quality of Life Scale for Patients with Schizophrenia | 1 year
  The Quality of Life Scale for Patients with Schizophrenia is an interviewer-administered tool assessed through a semi-structured interview. It consists of 4 subscales-interpersonal relationships, occupational role, psychological symptoms, and use of daily objects and activities-and includes a total of 21 items. Higher scores indicate better functioning. The scale's Cronbach's alpha reliability coefficient is reported as 0.80.

CONTACTS AND LOCATIONS:
Locations (1):
- ERZURUM, Erzurum, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No